CLINICAL TRIAL: NCT03246438
Title: Choice Architecture and Mailed Outreach for Colorectal Cancer Screening
Brief Title: Choice Architecture and Colorectal Cancer Screening Outreach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 827818
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Cancer of Colon
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Colonoscopy only outreach and follow-up
  Interventions: Behavioral: Colonoscopy only
- Sequential Choice (Experimental): Colonoscopy outreach + mailed FIT follow-up
  Interventions: Behavioral: Colonoscopy outreach + mailed FIT follow-up
- Active Choice (Experimental): Colonoscopy + mailed FIT outreach and follow-up
  Interventions: Behavioral: Colonoscopy + Mailed FIT outreach and follow-up

INTERVENTIONS:
Behavioral: Colonoscopy only — Subjects will receive a mailed communication describing the importance of colorectal cancer screening with the option to schedule a colonoscopy through a VIP direct scheduling phone line. Subjects not scheduled after 4 weeks will receive a reminder letter to schedule colonoscopy.
  Other Names: Control
  Arms: Control
Behavioral: Colonoscopy outreach + mailed FIT follow-up — Subjects will receive a mailed communication describing the importance of colorectal cancer screening with the option to schedule a colonoscopy through a VIP direct scheduling phone line. Subjects not scheduled after 4 weeks will receive a reminder letter to either schedule colonoscopy or to complete the enclosed mailed FIT kit.
  Other Names: Sequential Choice
  Arms: Sequential Choice
Behavioral: Colonoscopy + Mailed FIT outreach and follow-up — Subjects will receive a mailed communication describing the importance of colorectal cancer screening with the option to schedule a colonoscopy through a VIP direct scheduling phone line OR complete the enclosed mailed FIT kit. Subjects who have not completed FIT or scheduled colonoscopy within 4 weeks will be receive a reminder letter to either schedule colonoscopy or complete the mailed FIT kit previously sent.
  Other Names: Active Choice
  Arms: Active Choice

SUMMARY:
This pilot study is a 3-arm randomized control trial assessing the effectiveness of sequential or active choice in CRC (colorectal cancer) screening outreach vs. colonoscopy outreach only, in patients between 50-74 years old, who have received care at the University City or Valley Forge CCA (Community Care Associates) practices, are due for screening, and are asymptomatic for CRC. The three arms are: Arm 1: Direct schedule colonoscopy (Control), Arm 2: Direct schedule colonoscopy followed by mailed FIT(Fecal Immunochemical Test) (Sequential Choice), and Arm 3: Choice of direct schedule colonoscopy or mailed FIT (Active Choice).

DETAILED DESCRIPTION:
This pilot study is a 3-arm randomized control trial assessing the effectiveness of sequential or active choice in CRC screening outreach vs. colonoscopy outreach only. The investigators will randomize participants to one of three study arms:

Arm 1: Direct schedule colonoscopy (Control) Arm 2: Direct schedule colonoscopy followed by mailed FIT (Sequential Choice) Arm 3: Choice of direct schedule colonoscopy or mailed FIT (Active Choice).

ELIGIBILITY:
Inclusion Criteria:

* Between 50 and 74 years old
* Has a primary care provider who is a University City or Valley Forge Family Medicine provider
* Has had at least 2 office visits at either practice
* Is due for colorectal cancer screening
* Is asymptomatic for CRC
* Subject's zip code is within the Philadelphia-Wilmington-Camden Metropolitan Statistical Area

Exclusion Criteria:

* Has had prior colonoscopy within 10 years, sigmoidoscopy within 5 years, or FOBT/FIT within twelve months of chart review (we will exclude patients who self-report any of the above procedures)
* Has a history of CRC or colonic polyps
* Has a history of GI cancer
* Has a history of confirmed Inflammatory Bowel Disease (IBD)
* has a history of colitis other than Crohns disease or ulcerative colitis)
* Has a first degree relative that has been diagnosed with CRC
* Has had a colectomy
* Has been diagnosed with Familial Adenomatous Polyposis (FAP)
* Has been diagnosed with Lynch Syndrome (i.e. HNPCC)
* Has iron-deficiency anemia
* Has a history of lower GI bleeding
* Has metastatic (Stage IV) blood or solid tumor cancer
* Has end stage renal disease
* Has cirrhosis
* Has heart failure
* Has dementia
* Has any other condition that, in the opinion of the investigator, excludes the patient from participating in this study

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
CRC screening completion | 4 months
  The percentage of participants who successfully complete FIT or colonoscopy

SECONDARY OUTCOMES:
Choice of screening test | 4 months
  The percentage of participants who choose either screening method (FIT vs. colonoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania; Chyke Doubeni, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehta SJ, Induru V, Santos D, Reitz C, McAuliffe T, Orellana C, Volpp KG, Asch DA, Doubeni CA. Effect of Sequential or Active Choice for Colorectal Cancer Screening Outreach: A Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e1910305. doi: 10.1001/jamanetworkopen.2019.10305. PMID 31469393